CLINICAL TRIAL: NCT01579461
Title: An Open Label Single Dose Study to Investigate the Effect of Mild and Moderate Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of YM178 Compared With Healthy Subjects
Brief Title: A Study to Investigate the Effect of Mirabegron (YM178) on Subjects With Mild or Moderate Hepatic Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-039; 2008-000210-77 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Pharmacokinetics; Healthy Subjects; Mild and Moderate Hepatic Impairment
Keywords: Pharmacokinetics; mirabegron; hepatic impairment; Phase 1
MeSH Terms: conditions — Lymphoma, Follicular | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- mild hepatic impairment (Experimental)
  Interventions: Drug: mirabegron
- moderate hepatic impairment (Experimental)
  Interventions: Drug: mirabegron
- healthy volunteers (matched with mild hepatic) (Experimental)
  Interventions: Drug: mirabegron
- healthy volunteers (matched with moderate hepatic) (Experimental)
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178

SUMMARY:
The study aims to investigate and compare the effect of Mirabegron (YM178) on subjects with mild and moderate hepatic impairment compared to healthy subjects.

DETAILED DESCRIPTION:
Healthy subjects and subjects with mild and moderate hepatic impairment are admitted on Day 1. Subjects receive a single oral dose of Mirabegron in the morning of Day 1 and will remain in the unit till Day 5 with outpatient visits on Days 6 and 7 for healthy subjects and Days 6, 7, 9 and 11 for subjects with hepatic impairment. Blood sampling for PK assessment will be up to 144 hrs post dose for healthy subjects and up to 240 hrs post dose for subjects with hepatic impairment. An additional blood sample was obtained for all subjects 4 hrs post dose for protein binding.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index more than or equal to 18.0 and less than 32.0 kg/m2 (men and women)
* Subject is genotyped as an extensive metabolizer for CYP2D6
* For subjects with mild/moderate hepatic impairment: Hepatic dysfunction scored as mild impairment ((between 5-6 in the Child-Pugh's classification) and moderate impairment (between 7-9 in the Child-Pugh's classification)
* Healthy subject with normal hepatic function

Exclusion Criteria:

* Known or suspected hypersensitivity to mirabegron or any components of the formulations used
* A marked prolongation at screening of QT/QTC interval demonstrated by a mean QTcF interval >450 ms for male subjects and a mean QTcF interval >470 ms for female subjects (based on 3 ECGs)
* Abnormal pulse rate and/or blood pressure measurements at the pre-study visit taken in triplicate by means of an automatic device, after subject has been resting in supine position for 5 min: •Pulse rate <40 or >90 bpm; Mean systolic blood pressure <90 or >160 mmHg; Mean diastolic blood pressure <40 or >95 mmHg
* Healthy subjects: use of any prescribed or OTC drugs (except paracetamol, with a maximum of 3g/day) in the 2 weeks prior to admission to the clinical unit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Assess the single dose pharmacokinetics of Mirabegron in healthy subjects compared to subjects with hepatic impairment | Day 1 - Day 11
  AUCinf and Cmax

SECONDARY OUTCOMES:
Safety assessed by incidence of adverse events, lab tests, physical exam, ECG and vital signs | Day 1 - End of Study (Up to Day 19)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- FNsP Bratislava, nemocnica akad. L. Dérera; Klinika pracovného lekárstva a toxikológie, Bratislava, Slovakia

REFERENCES:
- [Background] Dickinson J, Lewand M, Sawamoto T, Krauwinkel W, Schaddelee M, Keirns J, Kerbusch V, Moy S, Meijer J, Kowalski D, Morton R, Lasseter K, Riff D, Kupcova V, van Gelderen M. Effect of renal or hepatic impairment on the pharmacokinetics of mirabegron. Clin Drug Investig. 2013 Jan;33(1):11-23. doi: 10.1007/s40261-012-0031-3. PMID 23208320